CLINICAL TRIAL: NCT02088528
Title: The Ghana Primary Tube Versus Trabeculectomy Study
Acronym: GPTVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tema Christian Eye Center (Other)
Collaborators: International Glaucoma Association (Unknown); HCA International Foundation (Unknown)
Responsible Party: Principal Investigator, Alex Spratt, Principal Investigator, Tema Christian Eye Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCEC 044/13-14
Record Dates: First submitted 2014-03-11; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aurolab glaucoma drainage device (Active Comparator)
  Interventions: Device: Aurolab glaucoma drainage device
- Trabeculectomy with mitomycin-c (Active Comparator)
  Interventions: Procedure: Trabeculectomy with mitomycin-c

INTERVENTIONS:
Device: Aurolab glaucoma drainage device — Patients undergoing surgery will receive an implant
  Other Names: AADI
  Arms: Aurolab glaucoma drainage device
Procedure: Trabeculectomy with mitomycin-c — Trabeculectomy surgery augmented by application of mitomycin C (0.4 mg/ml) to the sclera in the region of the trabeculectomy site for a period of exactly 3 minutes.
  Arms: Trabeculectomy with mitomycin-c

SUMMARY:
Medical treatment of glaucoma in West Africa is often unsuccessful because of the cost of medications, disease severity and poor compliance. Surgical treatment is likely to be a more practical solution.

The purpose of this study is to compare the safety and efficacy of the Aurolab glaucoma drainage device against trabeculectomy with mitomycin-c in a prospective randomised surgical study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years, inclusive
* Open angle glaucoma. Including primary open angle glaucoma, pseudoexfoliative and pigmentary glaucoma
* Intraocular pressure 18 - 40 mmHg on maximal tolerated or maximal affordable medical therapy
* Informed consent given and consent form signed.

Exclusion Criteria:

* Unwilling or unable to give consent, unwilling to accept randomisation, or unable to return for scheduled protocol visits
* Pregnant or nursing women
* No light perception vision
* Previous incisional intraocular surgery, other than uncomplicated clear corneal cataract surgery
* Previous ocular laser in study eye
* Iris neovascularisation or proliferative retinopathy
* Primary angle closure or primary angle closure glaucoma
* Iridocorneal endothelial syndrome or anterior segment dysgenesis
* Epithelial or fibrous downgrowth
* Aphakia
* Chronic or recurrent uveitis
* Steroid-induced glaucoma
* Severe posterior blepharitis
* Unwilling to discontinue contact lens use after surgery
* Previous cyclodestructive procedure
* Glaucoma secondary to penetrating keratoplasty, trauma, retinal disease/surgery or neovascular disease
* Conjunctival scarring from prior ocular surgery, trauma or cicatrizing disease precluding a superior trabeculectomy
* Need for glaucoma surgery combined with other ocular procedures (i.e. cataract surgery, penetrating keratoplasty, or retinal surgery) or anticipated need for urgent additional ocular surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2014-03; Primary Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in intraocular pressure | 3 months, 6 months, 1 year, 18 months, 2 years, 2½ years, 3 years, 3½ years, 4 years, 4½ years, 5 years

SECONDARY OUTCOMES:
Complication rates | 1 day, 1 week, 1 month, 3 months, 6 months, 1 year, 18 months, 2 years, 2½ years, 3 years, 3½ years, 4 years, 4½ years, 5 years
Visual acuity | 1 day, 1 week, 1 month, 3 months, 6 months, 1 year, 18 months, 2 years, 2½ years, 3 years, 3½ years, 4 years, 4½ years, 5 years
Visual field | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Reoperation for glaucoma | 1 day, 1 week, 1 month, 3 months, 6 months, 1 year, 18 months, 2 years, 2½ years, 3 years, 3½ years, 4 years, 4½ years, 5 years
Supplemental medical therapy | 1 day, 1 week, 1 month, 3 months, 6 months, 1 year, 18 months, 2 years, 2½ years, 3 years, 3½ years, 4 years, 4½ years, 5 years
Quality of life | 1 week, 1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years

OTHER OUTCOMES:
Patient satisfaction with communications by text message | 1 week, 1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Spratt, MBBCh FRCOphth, Principal Investigator — Tema Christian Eye Center; Keith Barton, MBBCh MD FRCP FRCOphth, Study Chair — Moorfields Eye Hospital NHS Foundation Trust; Donald L Budenz, MD MPH, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- Tema Christian Eye Center, Tema, Ghana

REFERENCES:
- See also: Related Info — http://www.gptvt.com